CLINICAL TRIAL: NCT03542838
Title: Phase 1b Double-blind Study to Assess the Safety, Tolerability and Preliminary Efficacy of Intra-articular Administration of Resiniferatoxin Versus Placebo for the Treatment of Pain Due to Moderate to Severe Osteoarthritis of the Knee
Brief Title: Study of Resiniferatoxin for Knee Pain in Moderate to Severe Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTVA OA-001
Record Dates: First submitted 2018-05-07; First posted 2018-05-31 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee; Pain, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — resiniferatoxin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Except for the sentinel subject, the treatment assigned to each subject in the dose-escalation cohorts is blinded to the subject, investigators, and sponsor study team. The sentinel subject, the first subject in each dose-escalation cohort, is dosed with resiniferatoxin in an open-label fashion. Subjects in the dose-escalation cohorts who received placebo may receive resiniferatoxin in an open-label fashion after unblinding. All subjects in the dose-expansion cohorts are dosed with resiniferatoxin in an open-label fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resiniferatoxin (Experimental): Resiniferatoxin is administered as a one-time dose, intra-articularly at a dose level of 5ug, 12.5ug, 20ug, 25ug, or 30ug.
  Interventions: Drug: Resiniferatoxin
- Saline (Placebo Comparator): Saline is administered as a one-time dose, intra-articularly.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Resiniferatoxin — Resiniferatoxin is a compound purified from natural sources.
  Other Names: RTX
  Arms: Resiniferatoxin
Drug: Saline — Saline is a normal physiological solution
  Other Names: Normal saline
  Arms: Saline

SUMMARY:
This study evaluates the safety of resiniferatoxin in patients with moderate to severe knee pain due to osteoarthritis.

DETAILED DESCRIPTION:
This study is to evaluate the safety of resiniferatoxin administered intra-articularly to subjects with moderate to severe knee pain due to osteoarthritis (OA). It is also to assess the preliminary efficacy of resiniferatoxin to relieve knee pain when walking.

ELIGIBILITY:
Inclusion criteria:

1. Age: 35 years to 85 years
2. Diagnosis of moderate to severe pain due to OA: Moderate to severe osteoarthritis, based on American College of Rheumatology (ACR) criteria
3. BMI < 45 kg/m2
4. Pain in the target knee has been treated with at least 2 analgesic agents, including at least one NSAID
5. Prior failure in at least two prior analgesic agents (at least one NSAID)
6. Willing to abstain from other intra-articular treatments of the knee or any knee surgery for at least 24 weeks after treatment
7. Ability to comply with the study and give informed consent
8. If on an opioid medication, stable dose for at least 4 weeks prior to injection with no increase in dose leading up to study injection
9. If on NSAIDs, be on a stable analgesic regimen for at least 4 weeks prior to injection
10. If on pain regimens other than opioid medication or NSAIDs, be on a stable regimen for at least 30 days
11. Is in good general health and is considered to have a physical status that is American Society of Anesthesiologists (ASA) category ≤ 3
12. Able to comply with study procedures, including the recording of daily questionnaires

Exclusion Criteria:

1. Has evidence or history of a coagulopathy or hemostasis problem at Screening or Baseline (Day 1)
2. Treatment knee injections with corticosteroids within 30 days or hyaluronic acid within 3 months prior to the procedure
3. If on opioid analgesics, an upper limit of 30 mg/day of oral morphine sulfate, 20 mg/day of oxycodone, 30 mg/day of hydrocodone, or 300 mg/day of tramadol, or equivalent
4. Any of the following lab abnormalities within one week of the treatment day:

   * Platelet count <100,000 cells/mm3
   * Total neutrophil count <1500 cells/mm3
   * Serum creatinine ≥ 1.5 x ULN
   * Alanine aminotransferase (ALT) > 3.0 x ULN
   * Aspartate aminotransferase (AST) > 3.0 x ULN
   * Alkaline phosphatase > 2.0 ULN
   * Bilirubin > 1.5 x ULN
   * INR > 1.5 x ULN
   * Temperature ≥ 100.4°F or other evidence of an infection
5. Concurrent use of opioids for indications other than knee pain
6. History of substance abuse
7. Has an allergy or hypersensitivity to chili peppers, capsaicin, resiniferatoxin or radiographic contrast agents
8. Female subjects who are pregnant at Screening or are planning on becoming pregnant, or are currently breastfeeding
9. Subjects with any medical condition or comorbidities that could adversely impact study participation or safety, conduct of the study, or interfere with pain assessments
10. Subjects who have participated in a clinical study of an investigational drug within 4 half-lives of Screening or are scheduled to receive and investigational agent while participating in this study
11. Sensory peripheral neuropathy that is CTCAE Grade 2 or higher at Screening
12. Arterial or venous thrombi, myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within 12 months prior to Screening
13. Evidence or history of any hemorrhage or bleeding event that is higher than CTCAE Grade 1 within 4 weeks prior to injection.
14. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C. Positive tests for HIV-1 or -2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies.
15. Concurrent medical or arthritic conditions that could interfere with evaluation of the index knee joint including fibromyalgia, rheumatoid arthritis, or other inflammatory arthropathies affecting the knee joint
16. Subjects with significant pain in other joints may be excluded at the discretion of the investigator
17. Subject has undergone arthroscopic or open surgery to the knee within 6 months of the planned injection day
18. Subject has undergone replacement surgery of the treatment knee
19. Presence of surgical hardware or other foreign bodies in the treatment knee

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Safety measurement | baseline through week 52
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Improvement of knee pain when walking | baseline through week 52
  Improvement in pain score versus baseline using the WOMAC Osteoarthritis Index question A1 (pain on walking, 11-point numerical rating scale)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, MD, Study Director — Sorrento Therapeutics
Locations (4):
- United States (4):
  - Snibbe Orthopedics, Los Angeles, California
  - University of Miami/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Hermann Drive Surgical Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No